CLINICAL TRIAL: NCT01022684
Title: Correlation of Inflammatory Markers Such as LpPLA2,MCP-1 and hsCRP for Predicting Vascular Inflammation; Analysis With 18F-Fluorodeoxyglucose Positron Emission Tomography
Brief Title: Correlation Between Various Inflammatory Markers and Vascular Inflammation Measured by 18FDG-PET
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Kyung Mook Choi, Korea University
Other Study IDs: KOSEF20546
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2009-11

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; vascular inflammation; LpPLA2; hsCRP; MCP-1; 18FDG-PET
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy patients
  Interventions: Other: Cross section study

INTERVENTIONS:
Other: Cross section study — This is not intervention study. The purpose of the study is to examine the relationship between various inflammatory markers and PET imaging at the cross section setting

SUMMARY:
Vascular inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis. Various inflammatory markers such as LpPLA2,MCP-2 and hsCRP are well-known prognostic factors for the cardiovascular event.

18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques.Therefore, the purpose of the study is to demonstrate the correlation between various inflammatory markers and vascular inflammation detected by 18FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Diabetes
* Stage 2 hypertension (resting blood pressure, ≥160/100 mmHg)
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect inflammation such as NSIAD and statin

Ages: 20 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participatin who underwent a medical health check in the health promotion center in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Correlation between various inflammatory markers including LpPLA2,MCP-1 and hsCRP and vascular inflammation analyzed by 18FDG-PET | 12 weeks

SECONDARY OUTCOMES:
Correlation between various inflammatory markers and atherosclerosis measured by carotid intima media thickness | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD.PhD, Principal Investigator — Korea University
Locations (1):
- Hye Jin Yoo, Seoul, South Korea

REFERENCES:
- [Derived] Yang SJ, Kim S, Choi HY, Kim TN, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. High-sensitivity C-reactive protein in the low- and intermediate-Framingham risk score groups: analysis with 18F-fluorodeoxyglucose positron emission tomography. Int J Cardiol. 2013 Mar 10;163(3):277-281. doi: 10.1016/j.ijcard.2011.06.054. Epub 2011 Jun 29. PMID 21719129